CLINICAL TRIAL: NCT02829931
Title: Phase I Trial of Hypofractionated Stereotactic Irradiation (HFSRT) Combined With Nivolumab, Ipilimumab and Bevacizumab in Patients With Recurrent High Grade Gliomas
Brief Title: Hypofractionated Stereotactic Irradiation With Nivolumab, Ipilimumab and Bevacizumab in Patients With Recurrent High Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18661
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Malignant Glioma
Keywords: recurrent glioma; high grade glioma; head and neck disease; grade III glioma; grade IV glioma; radiation therapy
MeSH Terms: conditions — Glioma | interventions — Radiotherapy; Nivolumab; Bevacizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Safety Cohort: The first 6 participants will receive Hypofractionated Stereotactic Irradiation (HFSRT) followed by Ipilimumab + Nivolumab + Bevacizumab.
  Dose Expansion Cohort: All 26 participants will be treated with Hypofractionated Stereotactic Irradiation (HFSRT), followed by Ipilimumab + Nivolumab +Bevacizumab
  Interventions: Radiation: Hypofractionated Stereotactic Irradiation; Drug: Nivolumab; Drug: Bevacizumab; Drug: Ipilimumab

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Irradiation — Hypofractionated Stereotactic Irradiation (HFSRT) prior to nivolumab.
  Other Names: HFSRT; radiation therapy
Drug: Nivolumab — Nivolumab intravenously (IV): 240 mg every (q) 3 weeks x 4 months followed by 480 mg X 4 months.
  Other Names: OPDIVO
Drug: Bevacizumab — Bevacizumab intervenously (IV): 15 mg/kg every (q) 3 weeks when given with Ipilumumab and Nivolumab combination. Dose changed to 10mg/kg every 2 weeks when given with Nivolumab only.
  Other Names: Avastin
Drug: Ipilimumab — Ipilimumab 1mg/kg intervenously (IV) 200 mg (5 mg/mL) every (q) 3 weeks for 4 months.
  Other Names: Yervoy

SUMMARY:
The main purpose of this study is to evaluate the safety, and tolerability of nivolumab, ipilimumab, and bevacizumab given in combination with hypofractionated stereotactic re-irradiation of recurrent high grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of World Health Organization (WHO) Grade III or IV malignant glioma.
* Documented recurrence by diagnostic biopsy or contrast enhanced magnetic resonance imaging (MRI) performed within 28 days of entry in to the trial as per Response Assessment in Neuro-Oncology (RANO) criteria.
* Maximum diameter of enhancing tumor (target lesion) should be ≤ 4 cm.
* An interval of at least 6 months after the end of prior radiation therapy is required unless there is a new recurrence outside of the previous radiotherapy treatment field.
* Previous first line treatment with at least standard dose of radiotherapy (total dose ≥ 54 Gy) and temozolomide or Procarbazine, Lomustine, and Vincristine (PCV) for high grade glioma.
* An interval of ≥ 4 weeks since surgical resection prior to start of study treatment.
* An interval of ≥ 4 weeks after the last administration of any investigational agent, bevacizumab, or prior cytotoxic therapy.
* ≥18 years of age on day of signing informed consent.
* Karnofsky performance status of 70 or higher.
* Demonstrate adequate organ function. All screening labs should be performed within 28 days of treatment initiation.
* Resting baseline O2 saturation by pulse oximetry of ≥ 92% at rest.
* Must have recovered from the toxic effects of prior therapies (≤ Grade 1).
* Willing and able to provide written informed consent for the trial.
* Life expectancy ≥ 12 weeks
* Women of childbearing potential (WOCBP) should have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. WOCBP should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication.
* Males should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.

Exclusion Criteria:

* Has more than three recurrences of high grade glioma. Previous recurrences of low grade glioma is not considered.
* Has received re-radiation to recurrent disease (other than standard frontline adjuvant radiation therapy).
* Recurrent tumors near the brainstem and optic chiasm must not have received prior radiation therapy.
* Has infratentorial, or leptomeningeal evidence of recurrent disease.
* Has recurrent or persistent tumor (enhancing area) greater than 4 cm in maximum diameter.
* Has prior treatment with Gliadel unless it was administered as first line treatment and at least 3 months prior to study treatment.
* Is unable (due to existent medical condition) or unwilling to have a contrast enhanced MRI of brain.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Low doses of steroid therapy (dexamethasone 2mg/day or ≤ 10 mg/day prednisone equivalents) is allowed.
* Has had a prior chemotherapy, targeted small molecule therapy, or monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. This does not include lymphopenia.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Potential participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Potential participants that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Potential participants with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Had major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of treatment on study.
* Requires escalating or chronic supraphysiologic doses of corticosteroids (>2 mg dexamethasone or > 10 mg/day prednisone equivalents) at the start day of treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator.
* Has prior history of uncontrolled hypertension, hypertensive crisis or hypertensive encephalopathy.
* Has history of non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to entry into the trial.
* Has history of gastrointestinal bleeding or any other hemorrhage/bleeding event ≥ grade 3 (CTCAE, v. 4) within 30 days prior to entry in to the trial.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-angiogenic agent such as bevacizumab, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C Virus (HCV) (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events | Up to 24 months
  Safety and tolerability of nivolumab, given in combination with hypofractionated stereotactic re-irradiation of recurrent high grade gliomas.

SECONDARY OUTCOMES:
Response Rate | Up to 36 months
  All participants will receive efficacy assessments with brain MRI at time points specified in Trial Flow Chart. Cases of suspected radiologic disease progression will be confirmed by an MRI performed approximately 8 weeks after the initial radiological assessment of progression. Immunotherapy Response Assessment in Neuro-Oncology (iRANO) and Response Assessment Criteria for High-Grade Gliomas (RANO Criteria) will be used for assessing the response to study treatment.
Overall Survival (OS) Rate at 6 Months | 6 months
  OS, utilizing 95% confidence interval (95%CI).
Overall Survival (OS) Rate at 9 Months | 9 months
  OS, utilizing 95% confidence interval (95%CI).

CONTACTS AND LOCATIONS:
Overall Officials: Solmaz Sahebjam, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/